CLINICAL TRIAL: NCT00836966
Title: Diagnostic Utility of Cytokine Biomarkers in the Evaluation of Acute Knee Pain
Brief Title: Sampling Biomarkers in Meniscus Injury to the Knee
Status: Completed | Type: Observational
Sponsor: Scuderi, Gaetano J., M.D. (Other)
Collaborators: Stanford University (Other)
Responsible Party: Gaetano J Scuderi, MD, Stanford University
Other Study IDs: Scu.Cyt.001
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Cartilage Diseases
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saline lavage from joint space
Oversight: Data Monitoring Committee: No

SUMMARY:
The diagnosis of clinically-significant meniscal tears of the knee remains challenging, and it is unknown why only some injuries become painful. The limitations of diagnostic magnetic resonance imaging result in arthroscopy that is not always beneficial. Elucidation of biochemical pathways underlying pain in this condition may aid patient selection for surgery and provide pharmacotherapeutic targets. Cytokines may be involved in pain following meniscus injury and diagnostic cytokine assay may help physicians differentiate patients that may benefit from arthroscopy from those that may not.

DETAILED DESCRIPTION:
Lavage of the operative and contralateral knee for comparison was performed under anesthesia prior to arthroscopy by the infusion of sterile saline into the knee joint followed by the immediate withdrawal into the syringe. Sixteen asymptomatic control subjects also contributed knee samples. The concentrations of 17 inflammatory cytokines/chemokines were measured using a multiplexed immunoassay panel. Pre-operative magnetic resonance imaging findings and cytokine assay results were compared to "gold-standard" intraoperative findings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with knee pain < 6 months with acute onset who had failed conservative treatment and elected for arthroscopic management. Indications for surgery included the presence of mechanical symptoms on history, a physical examination positive for McMurray's maneuver or joint line tenderness or both32, absence of severe joint space narrowing on plain radiography1 33, and the presence of grade III signal changes on MRI35 in an anatomic location consistent with the history and physical examination.

Exclusion Criteria:

* Less than 18 years old.
* Recent (within three months) intra-articular corticosteroid injection and past or current medical history of autoimmune disease (i.e. rheumatoid arthritis).
* In addition, no patients involved in a worker's compensation claim or personal injury litigation were enrolled in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 68 patients with knee pain < 6 months with either acute or insidious onset who failed conservative management and elected arthroscopy. Adult volunteers with no history of knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano J Scuderi, MD, Principal Investigator — Stanford University